CLINICAL TRIAL: NCT02562456
Title: Difference of Cost-efficacy Between Atraumatic Restoration Treatment (ART) and Composite Resin Restorations in Primary Molars: A Randomized Clinical Trial
Brief Title: Cost-efficacy Between ART and Composite Resin Restorations in Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associate Professor of Pediatric Dentistry Department, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECART
Record Dates: First submitted 2015-09-21; First posted 2015-09-29 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Dental Caries
Keywords: Dental Atraumatic Restorative Treatment; Composite Resins; Primary Teeth; Clinical Efficacy; Cost Analysis
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Treatment (Active Comparator): Occlusal and occlusoproximal composite resin restorations in primary molars (rubber dam isolation + Adhesive system + composite resin Filtek z350)
  Interventions: Procedure: Conventional Treatment
- ART using Fuji IX (Experimental): Occlusal and occlusoproximal ART restorations in primary molars with GIC Fuji IX
  Interventions: Procedure: ART using Fuji IX

INTERVENTIONS:
Procedure: ART using Fuji IX — Occlusal and occlusoproximal ART restorations in primary molars using the high viscosity GIC Fuji IX will be performed under relative isolation. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with GIC. After the press-finger technique, the excess of material will be removed and occlusion will be checked. For occlusoproximal restoration, an adapted matrix strip with a wooden wedge will be used to assure appropriate contour.
  Arms: ART using Fuji IX
Procedure: Conventional Treatment — Occlusal and occlusoproximal composite resin restorations in primary molars using the Scotchbond Multi-purpose adhesive system and the Filtek Z-350 composite resin wil be performed. Local anesthesia will be used. Absolute isolation will be performed using rubber dam and clamp. Removal of unsupported enamel will be performed using a round bur. Infected carious tissue will be removed with hand instruments. The cavity will be etched using 37% phosphoric acid for 15 seconds followed by rising and drying for the same amount of time. The cavity will be restored with composite resin. Occlusion will be checked. an adapted matrix strip with a wooden wedge will be used to assure appropriate contour.
  Arms: Conventional Treatment

SUMMARY:
The aim of this randomized clinical trial study is to compare the longevity of Atraumatic Restorative Treatment (ART) using high viscosity GIC and Conventional Treatment using composite resin under rubber dam isolation and local anesthesia (CT) in primary molars. As secondary outcomes, cost-efficacy, self-reported discomfort and cooperation will also be tested. Children aging between 3 to 6 years old presenting at least one occlusal and/or occlusoproximal cavity will be randomly assigned to one of two groups according to the dental treatment: ART (experimental group) or CT (control group). The dental treatment will be performed at a dental care trailer located in a Public School in Barueri (São Paulo, Brazil). The unit of analysis for randomization will be the child. A number of 204 teeth presenting occlusal cavities and 240 teeth presenting occlusoproximal cavities were set after sample size calculation. The primary outcome will be the restorations' longevity, which will be assessed after 6, 12, 18 and 24 months by two evaluators through clinical examination according to Frencken et al. (1998) criteria for occlusal restorations and Roeleveld et al. (2006) criteria for occlusoproximal restorations. The time spent during the dental treatment and all materials used will be considered for estimating the cost-efficacy of each treatment. The individual's discomfort will be also measured after each dental procedure using the Facial Scale of Wong-Baker. Cooperation will be assessed by the operator using a 5-point scale.

DETAILED DESCRIPTION:
Research setting

The study will be performed in a dental care trailer which simulated a regular dental office and it is located inside a public school of the city Barueri (São Paulo, Brazil).

Sample size calculation

For sample size calculation, data regarding longevity of CT in occlusal and occlusoproximal restorations after 2 years were extracted from the literature as 86% for occlusal and 60% for occlusoproximal restorations. A difference of 15% and 20% between the longevity of CT and ART was set as non-inferiority limit. Considering the level of significance as 5%, power as 80% and adding 40% due to the study design (cluster per child), a number of 204 occlusal restorations and 240 occlusoproximal restorations will be needed.

Randomization

The child will be the unit of randomization which means that all eligible teeth of a participant will be treated according the same restorative approach. Randomization list will be obtained using blocks of 4, 6 and 8 generated by software Sealed Envelope Ltd. Opaque, sealed and sequentially numbered envelopes will be used for randomizing all participants immediately before restorative treatments' beginning.

Allocation concealment

To assure allocation concealment, the participant will be randomized immediately before the treatment. When two or more cavities is available, preventing the finalization of the treatment in only one session, breach of allocation concealment will be signalized in the participants' record.

Blinding

Due to differences between the techniques, it will be not possible to blind operators, participants and evaluators.

Operators

All operators will be masters or PhD students from the Pediatric Dentistry Department, Faculty of Dentistry, University of São Paulo, previously trained. All procedures will be performed with the assistance of a dental student previously trained to manipulate all restorative materials.

ELIGIBILITY:
Inclusion Criteria:

* Children aging between 3 and 6 years
* presenting good health conditions
* whose parents or legal guardians accept and sign the consent form
* with at least one occlusal or occlusal proximal caries lesion in primary molars
* only occlusal and/or occlusal-proximal surfaces with caries lesions with dentin involvement

Exclusion Criteria:

* severe behavioral issues
* presence of fistula or abscess near the selected tooth
* presence of pulp exposure in the selected tooth
* presence of mobility in the selected tooth

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 428 (Estimated)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2019-12-10 (Estimated)

PRIMARY OUTCOMES:
The restoration survival | Every 6 months up to 24 months.
  The treatments will be classified as successful when they present a clinical satisfactory aspect. Otherwise, "minor failures" will be analyzed. "Minor failures" are those in which there is a defect in the restoration/crown, but it does not interfere with the tooth health.

SECONDARY OUTCOMES:
Cost-efficacy assessment | Through study completion, an average of 24 months
  Treatment costs = professional costs + procedure costs.
  * Professional cost: the time spent in each session will be converted in hours and multiplied not only by the medium income of the dentist per hour added 40% of dangerousness but also by the medium income of a dental assistant added 20% of insalubrity
  * Procedure cost: variable cost (equipment & instruments depreciation and electricity) and and materials cost. To calculate the equipments' and instruments' depreciation, we will consider their price, the lifespan of 5 and 3 years respectively and a monthly use of 160 hours. To calculate materials' costs, all materials used in each procedure will have their specifications and quantity registered. Prices will be inferences from the market value converted in US Dollars obtained by the medium of the values from different places that commercialized the referred products.
  If the restorative treatment requires repairs, the additional cost of it will also be considered.
Child self-reported discomfort | Immediately after treatment
  The acceptability of each type of treatment will be evaluated using the Facial scale of Wong-Baker (Wong; Baker, 1998). This scale indicates the discomfort of an individual who has to choose among six faces, each one expressing different facial countenance. The first image is a smiling happy face, indicating no discomfort, followed by gradually less cheerful expressions, up to the last one which is a very sad face covered by tears, indicating great discomfort. The participant will be asked to choose the face that is more similar to how he or she felt during the treatment. This answer should be given solely by the child, which means, no parental or professional interferences. The facial scale of Wong-Baker will be applied right after the end of each restorative treatment session.
Cooperation | Immediately after treatment
  Cooperation will be evaluated by the operator immediately after the end of the treatment using a 5-point scale: 1- Good behaviour, 2- Reasonable behaviour, 3- Indiferent, 4- Bad behaviour, 5- Really bad behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Complexo Educacional Carlos Osmarinho de Lima - Trailer USP, Barueri, São Paulo, Brazil

REFERENCES:
- [Derived] Ladewig NM, Sahiara CS, Yoshioka L, Olegario IC, Floriano I, Tedesco TK, Mendes FM, Braga MM, Raggio DP. Efficacy of conventional treatment with composite resin and atraumatic restorative treatment in posterior primary teeth: study protocol for a randomised controlled trial. BMJ Open. 2017 Jul 10;7(7):e015542. doi: 10.1136/bmjopen-2016-015542. PMID 28698331